CLINICAL TRIAL: NCT04841434
Title: An Open Label, Phase I/II Study to Investigate the Use of VORAXAZE™ As Intended Intervention in Patients with Central Nervous System Lymphoma and with Impaired Renal Function Being Treated with High-dose Methotrexate
Brief Title: A Phase I/II Study to Investigate the Use of VORAXAZE™ As Intended Intervention in Patients with CNSL
Acronym: VALIDATE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Schwartz, PD Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-Lymphoma-Vorax-1
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: CNS Lymphoma
Keywords: impaired renal function
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Dose escalation will be performed using three dose levels of MTX.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): Patients will receive up to 6 cycles of HD-MTX Treatment Dose escalation will be performed using three dose levels of MTX: 3.0 g/m2, 3.5 g/m2, 4.0 g/m2
  Interventions: Drug: Voraxaze Injectable Product

INTERVENTIONS:
Drug: Voraxaze Injectable Product — High-dose Methotrexat Infusion: MTX is given at a dose according to the allocated dose level cohort as a 4-hour IV infusion. HD-MTX cycles (up to 6) should be repeated every 14 days, provided that the patient has recovered (i.e., hematopoietic reconstitution) between cycles. A delay of up to 28 days between cycles is permitted in order to allow patients to recover from the preceding dose of MTX. In patients with a decline of the GFR to <40 mL/min, or in the case of decreased GFR, the decrease is >50% compared with the pretreatment value, treatment will be terminated. At the start of Cycle 3 the dose of MTX can be escalated to the next level if MTX has been well-tolerated according to the criteria described under dose escalation. Voraxaze: 2000 Units in patients weighing ≤100kg and at least 20 Units per kg body weight in patients weighing >100kg is given in each HD-MTX cycle as a slow IV injection at 24 hours (+/- 2 hours) after the start of HD-MTX infusion.
  Other Names: High-dose Methotrexat Infusion

SUMMARY:
This phase I-II trial is intented to demonstrate tolerability (i.e. absence of severe non-hematological toxicity) and efficacy of intended intervention with repeated doses of Voraxaze, in addition to leucovorin (LV), in patients with renal impairment or renal failure during previous HD-MTX therapy.

Patients will receive up to 6 cycles of HD-MTX treatment with 14 days between cycles (a maximum delay of 28 days is permitted in order to allow time for a patient to recover from the previous cycle).

DETAILED DESCRIPTION:
MTX is used either alone or as part of a combined chemotherapy protocol either in standard or high doses in the treatment of a range of cancers and other diseases.

Dose escalation will be performed using three dose levels of MTX:

Level 1: 3.0 g/m2 Level 2: 3.5 g/m2 Level 3: 4.0 g/m2 Up to 6 patients will be treated at each dose level; each will receive a maximum of 6 cycles of treatment. The dose may be increased in Cycle 3 in individual patients to the next level, if renal function is adequate (GFR ≥ 40 mL/min, or in the case of decreased GFR, the decrease is <10% compared with the pre-treatment value), and absence of grade 3 or 4 non-hematological toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary CNSL (PCNSL or SCNSL) confirmed by histology or cytology.
* Renal insufficiency defined as a glomerular filtration rate (GFR, assessed by CKD-EPI or MDRD equation) of 40-80 mL/min or patients with a GFR >80mL/min who have experienced renal failure, defined as doubling of the serum creatinine compared to the baseline value during a previous HD-MTX treatment.
* Age ≥ 18 years (male or female).
* Life expectancy >3 months.
* Adequate organ function (i.e., bone marrow, liver, lungs) allowing intensive chemotherapy with MTX.
* Adequate clinical pathology values:
* Absolute neutrophil count ≥1.0 x 109/L, hemoglobin ≥9mg/dL (transfusion allowed), platelets ≥100 x 109/L.
* Total bilirubin ≤1.5x the upper limit of normal except for patients with known Gilbert syndrome.
* Alanine amino-transferase (ALT) and aspartate amino-transferase (AST) ≤2x the upper limit of normal.
* Alkaline phosphatase ≤2x the upper limit of normal.
* Prothrombin time within the normal range for the institution.
* Signed informed consent by the patient or legal representative prior to start of any study specific procedure.
* Females of childbearing potential and males must be willing and able to use an adequate method of contraception to avoid pregnancy for the duration of the study in such a manner that the risk of pregnancy is minimized. Acceptable contraceptives include intra-uterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.

Exclusion Criteria:

* Ongoing or expected need for therapy with drugs interfering with MTX-clearance (i.e., beta-lactam antibiotics, NSAIDs, probenicid, salicylates, sulphonamides) or other nephrotoxic drugs.
* Prior brain radiotherapy within 28 days of first dose of the study drug.
* Concurrent illness interfering with hydration (i.e., relevant congestive heart failure, SIADH syndrome).
* Relevant third space (i.e., pleural effusion, ascites, extended edema) precluding HD-MTX treatment.
* Obesity (body mass index >30 kg/m2).
* Uncontrolled diabetes.
* Active hepatitis.
* HIV-infection.
* Pregnant or lactating woman.
* Participation in any other clinical trial either 1 month prior to or during this study.
* Previous intolerance to any of the drugs used in this study (i.e., MTX, LV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of Voraxaze | 1 year
  absence of severe non-hematological toxicity
Efficacy of Voraxaze | 1 year
  immediate and sustained reduction in plasma MTX concentration

SECONDARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | 1 year
  appearance of DLTs for each dose level of MTX
Anti-glucarpidase antibodies | at screening, prior to the MTX infusion at each treatment cycle and on day 28 of the last cycle
  presence of antibodies to glucarpidase
MTX toxicities | 1 year
  incidence and severity of hematological toxicities and stomatitis after each cycle of HD-MTX treatment and renal function before each cycle of HD-MTX treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Benjamin Franklin (CBF), Berlin, Germany